CLINICAL TRIAL: NCT06196580
Title: A Clinical Study Evaluating the Pharmacokinetic Effects of SHR4640 on Repaglinide and Midazolam in Healthy Subjects and the Impact of SHR4640 on QT Interval
Brief Title: PK Effects of SHR4640 on Repaglinide and Midazolam, and the Impact of SHR4640 on QT Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR4640-113
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gout and Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — repaglinide; Midazolam; ruzinurad

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, double blind, three-period, and three-group parallel design trial, consisting of three groups (group A、 group B and placebo group).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR4640 group A (Experimental)
  Interventions: Drug: repaglinide; midazolam; SHR4640
- SHR4640 group B (Experimental)
  Interventions: Drug: repaglinide; midazolam; SHR4640; SHR4640 placebo
- SHR4640 Placebo (Placebo Comparator)
  Interventions: Drug: repaglinide; midazolam; SHR4640 placebo

INTERVENTIONS:
Drug: repaglinide; midazolam; SHR4640 — repaglinide; midazolam; SHR4640
  Arms: SHR4640 group A
Drug: repaglinide; midazolam; SHR4640; SHR4640 placebo — repaglinide; midazolam; SHR4640; SHR4640 placebo
  Arms: SHR4640 group B
Drug: repaglinide; midazolam; SHR4640 placebo — repaglinide; midazolam; SHR4640 placebo
  Arms: SHR4640 Placebo

SUMMARY:
The purpose of this study is to evaluate the PK effects of SHR4640 tablets on repaglinide and midazolam, as well as the effects of SHR4640 tablets on the QT interval in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the trial-related activities, and be able to understand the procedures and methods of the trial, and are willing to strictly comply with the clinical trial protocol to complete the trial;
2. Aged 18 to 45 years old (both ends included, subject to the time of signing the informed consent form), male or female;
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 19-26 kg/m2 (both ends included);
4. No fertility plan and agree to take non-drug high-efficiency contraceptive measures (see appendix 1 for details) within 28 days from signing the informed consent form to the last administration of the trial drug, and no plans for sperm donation or egg donation.

Exclusion Criteria:

1. Individuals who have a history of smoking within the 3 months before signing the informed consent form (average daily smoking>5 cigarettes) or who cannot stop using any tobacco products during the study period;
2. The average daily intake of alcohol in the three months before signing the informed consent is more than 7 g for women (about 200 ml beer, 70 ml wine or 22 ml low-alcohol liquor) and 14 g for men (about 400 ml beer, 140 ml wine or 45 ml low-alcohol liquor); Those who cannot abstain from alcohol during the trial;
3. Within the first 7 days of randomization, consumed any beverage or food containing grapefruit; Or have eaten any beverages or foods containing methylxanthines, such as coffee, tea, cola, chocolate, etc., within the previous 2 days at random;
4. Allergic constitution, or allergic or suspected allergic to SHR4640 tablets, repaglinide or midazolam;
5. Drug abusers, or those who have positive urinary abuse during screening;
6. any history of severe clinical disease or conditions that the researcher believes may affect the results of the trial, including but not limited to the history of circulatory, endocrine, nervous, digestive, urinary, or blood, immune, psychiatric, and metabolic diseases;
7. Patients with contraindication of repaglinide (type 1 diabetes, C-peptide negative diabetes patients, diabetes ketoacidosis patients with or without coma);
8. Patients with contraindications to midazolam (acute angle closure glaucoma, severe respiratory insufficiency, sleep apnea syndrome, myasthenia gravis, schizophrenia, and severe depressive state);
9. During screening, vital signs, physical examinations, laboratory tests, cardiac ultrasound, abdominal ultrasound, or chest imaging examinations indicate the presence of abnormalities that are clinically significant according to the judgment of the investigator;
10. When screening, ultrasound examination of the urinary system indicates the presence of stones or crystals in the urinary system;
11. Individuals with acute kidney injury before screening or random ;
12. Individuals with serum uric acid higher than 420 μmol/L at screening, , or a history of hyperuricemia and/or gout disease;
13. Individuals with QTcF>450 ms, PR interval>200 ms, QRS complex time limit>120 ms, or HR>100 bpm, or other abnormalities that were clinically significant as determined by the researcher;
14. Individuals with risk factors for torsade de pointe ventricular tachycardia, such as heart failure, hypokalemia, short QT syndrome, long QT syndrome, or a first-degree relatives family history of unexplained sudden death, drowning, or sudden infant death syndrome in young adulthood (≤ 40 years old);
15. Individuals with positive hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) antibodies, or syphilis antibodies during screening;
16. Individuals who have used any prescription drugs, over-the-counter drugs, herbal medicines, or dietary supplements within two weeks before randomization;
17. Systemic treatment with cytochrome P450 3A4 enzyme (CYP3A4), CYP2C8 inhibitor or inducer drugs used within the first 4 weeks of randomization ;
18. Individuals (excluding screening failures) who have participated in any other drug or medical device clinical trials within 3 months before randomization or within 5 half-lives of the trial drug (whichever is longer);
19. Individuals who have undergone any surgery within three months before randomization, or have not recovered after surgery, or plan to undergo surgery during the trial;
20. Individuals who have donated (or lost) blood within three months before randomization and the amount of blood donated (or lost) is ≥400 mL, or received blood transfusion;
21. According to the judgment of the researchers, subjects with conditions that affect drug absorption, distribution, metabolism, and excretion, or other factors that are not suitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: Cmax | Day 1 to Day 24
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: AUC0-t | Day 1 to Day 24
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: AUC0-inf | Day 1 to Day 24
QTcF corrected for baseline and placebo after oral administration of SHR4640 tablets（ ΔΔ QTcF） | Day 1 to Day 24

SECONDARY OUTCOMES:
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: Tmax | Day 1 to Day 24
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: t1/2 | Day 1 to Day 24
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: CL/F | Day 1 to Day 24
The plasma PK parameters of repaglinide, midazolam, and SHR4640 in combination: Vz/F | Day 1 to Day 24
PK parameters for oral SHR4640 tablets: Cmax | Day 1 to Day 24
PK parameters for oral SHR4640 tablets: AUC0-t | Day 1 to Day 24
PK parameters for oral SHR4640 tablets: Tmax | Day 1 to Day 24
Safety indicators: adverse events | Screening period up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng Y, Hu X, Pei Z, Zhang Z, Lin H, Feng S, Gao Z, Ma Y, Cao Z, Zhang Q, Zheng L, Zhang W, Shen K, Hu W. Evaluating the drug-drug interactions of SHR4640 on repaglinide and midazolam in healthy subjects. Expert Opin Drug Metab Toxicol. 2025 Jan-Feb;21(2):217-224. doi: 10.1080/17425255.2024.2428367. Epub 2024 Nov 14. PMID 39530130